CLINICAL TRIAL: NCT07003191
Title: Multicenter, Prospective, Observational Study of Metformin Hydrochloride and Empagliflozin Tablets (Enshuangping) in the Treatment of Type 2 Diabetes
Brief Title: Metformin Hydrochloride and Empagliflozin Tablets in the Treatment of Type 2 Diabetes
Status: Active, not recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Liaoning Health Industry Group Fushun Mining General Hospital (Unknown); Liaoning Health Industry Group Benxi Steel General Hospital (Unknown); Changsha Fourth Hospital (Other Government); Second Hospital of Shanxi Medical University (Other); The First People's Hospital of Kunshan (Other); Suzhou Ninth People's Hospital (Unknown); the First Affiliated Hospital of Anhui University of Science and Technology (Unknown); Mingguang People's Hospital (Unknown); the People's Hospital Longhua Shenzhen (Unknown); Afﬁliated Hospital of North Sichuan Medical College (Other); Yiyang County People's Hospital (Unknown); THE SECOND PEOPLE'S HOSPITAL, WUHU (Unknown); The First People's Hospital of Zhangjiagang (Unknown); Yixing People's Hospital (Other); Shijiazhuang People's Hospital (Other); Guiyang First People's Hospital (Unknown); Lanzhou University Second Hospital (Other); Tiefa Coal Industry Group General Hospital (Unknown); Southern Medical University Shenzhen Hospital (Unknown); The Second Hospital of Shijiazhuang (Unknown); Ningbo University Affiliated People's Hospital (Unknown); Dongyang People's Hospital (Other); Xiangyang Central Hospital (Other); Li Hui Li Hospital (Unknown); Nanning Second People's Hospital (Other); Hunan Provincial People's Hospital Ma Wang Dui Branch (Unknown); The Second Affiliated Hospital of Bengbu Medical College (Unknown); Ruyang County People's Hospital (Unknown); Kaifeng People's Hospital (Unknown); Dingzhou People's Hospital (Unknown); The Second People's Hospital of Changshu (Unknown); The Second Affiliated Hospital of Henan University of Science and Technology (Unknown); Dengzhou People's Hospital (Unknown); Taizhou First People's Hospital (Other); Red Cross Hospital, Hangzhou, China (Other); The First People's Hospital of Lin'an District (Unknown); China Resources Wugang General Hospital (Unknown); Yiwu Central Hospital (Other); The First People's Hospital of Jiashan County (Unknown); The First People's Hospital of Tongxiang City (Unknown); Shaoxing Central Hospital (Other); The First People's Hospital of Jiande City (Unknown); Beilun District People's Hospital (Unknown); Huantai County People's Hospital (Unknown); Fifth Affiliated Hospital of Guangzhou Medical University (Other); Sixth Hospital of Wuhan, Affiliated Hospital of Jianghan University (Other); The Affiliated Hospital of Shaanxi University of Chinese Medicine (Unknown); Zhangjiagang Traditional Chinese Medicine Hospital (Unknown)
Responsible Party: Principal Investigator, Yanbing Li, the director of the endocrinology department of the First Affiliated Hospital of Sun Yat-sen University, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: 2023-414
Record Dates: First submitted 2025-01-14; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Metformin Hydrochloride and Empagliflozin tables (Fixed-Dose Combination) — First-time treatment with Metformin Hydrochloride and Empagliflozin Tablets (metformin 500mg and empagliflozin 5mg per table) for at least 6 months

SUMMARY:
The main objective of this study is to evaluate the efficacy and safety of Metformin Hydrochloride and Empagliflozin Tablets in the treatment of type 2 diabetes in real-world clinical settings. A total of 2,600 type 2 diabetes patients were included in the study. The study observed the clinical glycemic control rate and adverse events over a period of at least 6 months from the prescription date to the end of continuous clinical follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, gender unrestricted;
2. Clinically diagnosed with type 2 diabetes;
3. First-time treatment with metformin and empagliflozin tablets;
4. HbA1c test results within 2 weeks prior to enrollment (rapid fingertip test results are acceptable);
5. Voluntary participation in the study and signing of informed consent form.

Exclusion Criteria:

1. Moderate to severe renal impairment (eGFR < 45 mL/min/1.73 m²), end-stage renal disease, or dialysis;
2. Acute or chronic metabolic acidosis, including diabetic ketoacidosis;
3. A history of severe allergy to empagliflozin, metformin, or any excipient in this product;
4. Currently or within the past month, participation in any other clinical trials;
5. Judged by the investigator to be unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient and inpatient patients
Sampling Method: Probability Sample
Enrollment: 2600 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
6-month clinical glycemic control rate | 6 months
  6-month clinical glycemic control rate (clinical control defined as HbA1c < 7.0%)

SECONDARY OUTCOMES:
Change in HbA1c from baseline | 12 months
  Change in HbA1c from baseline at 12 months
Change of β cell function | 12 months
  Change of β cell function at 12 months
Change of insulin sensitivity | 12 months
  Change of insulin sensitivity indicators at the end of study
Change of lipid profiles | 12 months
  Change of cholesterol, Triglyceride, high-density lipoprotein cholesterol (HDL-c) and low-density lipoprotein cholesterol (LDL-c) at the end of study
Change of body weight | 12 months
  Change of body weight at the end of study
Changes in echocardiographic indicators in type 2 diabetes patients with cardiovascular disease | 12 months
  Changes in echocardiographic indicators in type 2 diabetes patients with cardiovascular disease at the end of study
Change of blood pressure | 12 months
  Change of blood pressure at the end of study
Change of Quality of life assessment (EQ-5D) | 12 months
  Change of Quality of life assessment (EQ-5D) at the end of study
Incidence of adverse events | 12 months
  incidence of adverse events at the end of study

CONTACTS AND LOCATIONS:
Locations (1):
- Endocrinology Department, The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided